CLINICAL TRIAL: NCT00827216
Title: The Effect of Intravenous Erythromycin on Gastric Emptying in Patients Undergoing Rapid Sequence Intubation for Full Stomach - A Randomised, Placebo-controlled, Double-blind Study
Brief Title: The Effect of Intravenous Erythromycin on Gastric Emptying in Non-fasted Patients Before Emergency Total Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christoph Czarnetzki, Responsable Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAC 06-225; Swissmedic 2008 DR 2321 (Other: Swiss Agency for Therapeutic products)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Aspiration of Gastric Contents; Gastric Emptying
Keywords: Gastric emptying; emergency anesthesia; intravenous erythromycin
MeSH Terms: interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiologic saline (Placebo Comparator)
  Interventions: Drug: Placebo
- Erythromycine (Active Comparator)
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Placebo — For all patients, a standardised volume of 10 ml of the study drug (will be diluted in 90 ml NaCl 0.9% (total volume, 100 ml). Both, the study drug and the 90 ml NaCl bag will be prepared by the pharmacy. Using sterile syringes, the investigator will withdraw from this solution as many millilitres as necessary to obtain a volume that corresponds to 1 ml per kg bodyweight of the patient (i.e. for a 67 kg patient, 33 ml would be with withdrawn). Thus, the maximum volume that can be administered to a patient will be 100 ml (i.e. for a patient weighing ≥100 kg). Twenty minutes prior to the scheduled induction of anaesthesia, patients will receive their study drug solution as an intravenous infusion during 5 min.
  Arms: Physiologic saline
Drug: Erythromycin — For all patients, a standardised volume of 10 ml of the study drug (will be diluted in 90 ml NaCl 0.9% (total volume, 100 ml). Both, the study drug and the 90 ml NaCl bag will be prepared by the pharmacy. Using sterile syringes, the investigator will withdraw from this solution as many millilitres as necessary to obtain a volume that corresponds to 1 ml per kg bodyweight of the patient (i.e. for a 67 kg patient, 33 ml would be with withdrawn). Thus, the maximum volume that can be administered to a patient will be 100 ml (i.e. for a patient weighing ≥100 kg). Twenty minutes prior to the scheduled induction of anaesthesia, patients will receive their study drug solution as an intravenous infusion during 5 min. The regimen corresponds to 3 mg/kg of erythromycin.
  Other Names: Erythrocine®
  Arms: Erythromycine

SUMMARY:
In this study the investigators want to investigate the effect of a short intravenous infusion of Erythromycine on gastric emptying on patients considered "full stomac" and scheduled for Emergency operation. A gastroscopy will be done after intubation to controll the effect of the perfusion.

DETAILED DESCRIPTION:
Urgent or emergency surgery requires that fasting rules observed in elective settings are not respected. Patients who are anesthetized in such conditions are at risk for regurgitation and subsequent broncho-aspiration during induction of anaesthesia due to a full stomach; they often have ingested food or liquids before the injury, or they may have swallowed blood from oral or nasal injuries. Also, gastric emptying is delayed in these patients due to the stress of trauma.1 Already in 1946, Mendelson described the consequences of bronchoaspiration.2 Since, anaesthetists and emergency physicians have tried to avoid broncho-aspiration in emergency patients using premedication with pro-kinetic drugs (for instance, metoclopramide) or its complications with antacid substances, and through the use of a rapid sequence intubation procedure with cricoid pressure.

The incidence of aspiration is low, about 1.4 to 6 in 10'000 anaesthetics.3 About 6 in 100'000 anaesthetics will lead to a pulmonary complication due to broncho-aspiration and about 1 in 100'000 patients is likely to die due to aspiration.4 Thus, although episodes of broncho-aspiration are rare, efficacious prevention of this potentially lethal complication is important. One method to reduce the risk of broncho-aspiration during induction of anaesthesia is the pharmacological reduction of the gastric content (i.e. pre-treatment).

The primary objective of this study is to investigate the effect of a short intravenous infusion of erythromycin 3 mg/kg, administered 20 min before intubation on gastric emptying, in adults scheduled for rapid sequence intubation for full stomach. After intubation a gastroscopy will be done to see if there is any content in the stomac. The secondary objective is the assessment of tolerability and safety of a single intravenous dose of preoperative erythromycin in surgical patients.

This study is a single centre, stratified (according to emergency setting), randomised, placebo-controlled, double-blinded study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age ≥18 years, male or female.
* American Society of Anaesthesiology [ASA] status I, II or III.
* Non-starving patients presenting for surgery.
* Patients able to read and understand the information sheet and to sign the consent form.
* If the patient is female and of childbearing potential, she must have a negative pregnancy test

Exclusion Criteria:

* A history of allergy or hypersensitivity to erythromycin or other macrolides.
* Concomitant use of terfenadine, astemizole, cisapride, pimozid, cyclosporine, clarithromycine.
* Patient with acute intermittent porphyria.
* Acute or subacute necrosis of the liver, acute or subacute hepatitis, acute liver trauma
* Acute renal failure, acute glomerulonephritis, nephritic syndrome, chronic renal failure with electrolyte disorders, uremia
* Exacerbated asthma, exacerbated chronic obstructive lung disease, acute pulmonary infection
* Coronary heart disease (unstable angina, MI within the last 6 months), decompensated cardiac insufficiency, aortic aneurysm
* Polyneuropathy (for instance, due to diabetes mellitus)
* Patients with oesophageal and pharyngeal disease (i.e. oesophageal varices, oesophageal and pharyngeal cancer, Zenker's diverticulum).
* Status after gastric surgery, gastric bypass surgery, Nissen operation
* Patients with life threatening illness or injury needing immediate surgery
* Patients with moderate to severe head trauma (GCS on admission <13)
* Psychological or psychiatric disorders.
* Dementia or inability to understand the study protocol.
* Women who are pregnant or are breast feeding.
* Patient scheduled for ileus surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Immediately after intubation an upper GI endoscopy will be done. The following primary endpoint will be recorded: Stomach clear from any content: yes or no (dichotomous). | 10 minutes

SECONDARY OUTCOMES:
Acidity and Estimation of the volume of gastric content if stomach not empty (ml). | 10 minutes
Drug-related allergic reactions. | 30 minutes
Arrhythmia. | 30 minutes
Gastrointestinal cramps after study drug administration but before intubation. | 30 minutes
Nausea or vomiting after study drug administration but before intubation. | 30 minutes
Regurgitation with or without broncho-aspiration at induction. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, MBA, Principal Investigator — Division of Anesthesiology, University Hospital of Geneva; Martin R Tramer, MD, PhD, Study Chair — Division of Anesthesiology, University Hospital of Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Czarnetzki C, Elia N, Frossard JL, Giostra E, Spahr L, Waeber JL, Pavlovic G, Lysakowski C, Tramer MR. Erythromycin for Gastric Emptying in Patients Undergoing General Anesthesia for Emergency Surgery: A Randomized Clinical Trial. JAMA Surg. 2015 Aug;150(8):730-7. doi: 10.1001/jamasurg.2015.0306. PMID 26083537